CLINICAL TRIAL: NCT02655939
Title: Double Blind, Randomized, Multicentre, Placebo Controlled Study to Assess the Efficacy and Safety of Reflex Plus™ in Osteoarthritis
Brief Title: Study to Assess the Efficacy and Safety of Reflex Plus™ in Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Fullife Healthcare Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FZ/150603/RFX+/OA
Record Dates: First submitted 2015-12-02; First posted 2016-01-14 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis
Keywords: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Reflex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reflex Plus (Active Comparator): Reflex Plus TM, Sachets to be taken once in a day Before breakfast for the study duration
  Interventions: Dietary Supplement: Reflex Plus
- Placebo (Placebo Comparator): Placebo Sachets to be taken once in a day Before breakfast for the study duration
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Reflex Plus — Collagen Hydrolysate: 5g ,Rosehip aqueous extract 0.55g,
  Arms: Reflex Plus
Dietary Supplement: Placebo — Fructose,Orange flavor and sucralose
  Arms: Placebo

SUMMARY:
Reflex plus™ is a unique blend of Collagen Hydrolysate with Rosehip extract. The blend contains individual ingredients which have been widely studied for its effectiveness in osteoarthritis(OA). Collagen hydrolysate is accumulated in the cartilage and helps to repair the OA, related cartilaginous changes. Rosehip works in the anti-inflammatory pathway thus reducing the pain and inflammation of the joint.

The two open-label studies have showed the effectiveness of the investigational product on OA. The 2 studies did not show any specific safety concern to be considered. The study demonstrated the synergistic effect of CH and Rosehip extract from former in-vitro results in the formulation.

The supplement has been manufactured in GMP certified manufacturing units in Germany and India under strict quality control check. Hence, quality of the supplement and batch to batch consistency is well assured.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of Reflex Plus on osteoarthritis(OA) patients. The duration of the study is 12 / 24 weeks excluding the screening period of approximate 1 week. The test product being studied is Reflex Plus is composed of Collagen hydrolysate and Rosehip extract, it is a health supplement. It is expected to help in the building of cartilage for efficient joint functioning and relieving pain associated with arthritis It helps in cartilage protection and joint pain management.The primary endpoint of the study is the change in knee pain as measured by the WOMAC osteoarthritis (OA) index sum score between baseline and last visit in the comparison between IP and placebo.

ELIGIBILITY:
Inclusion Criteria

* Male and Female, aged ≥ 50 yrs and ≤ 70 yrs, with BMI<30.
* WOMAC pain score, between 8-16 on a scale of 0 to 20.
* Diagnosis confirmed of Gonarthrosis, by clinical and radiological means by Jaeger-Wirth score ≥2.
* Females to be included in the study should have reached menopause.
* Subjects willing to stop the restricted supplements and medications prior to inclusion in study and even during the study.
* Subjects using topical applications and rescue medication willing to stop the use 48 hours prior to all assessment.
* Subjects with Fasting blood glucose level ≤ 140 and Systolic blood pressure ≤ 160 mm of Hg and diastolic blood pressure ≤ 100 mm of hg.
* Subjects willing to adhere to protocol and complete subject diary.
* Patient willing and able to provide signed informed consent.

Exclusion Criteria

* Knee pain or functional impairment of the knee joint from causes other than osteoarthritis.
* Peripheral arterial occlusive disease
* Acute meniscus injuries
* Rheumatoid Arthritis
* Infection-associated arthritis
* Coxarthrosis
* Bony injuries of lower extremities(e.g. femoral neck fracture) in the last 12 months

Herniated Spinal Disc

* Any other severe organic and/or systemic diseases (e.g. renal, hepatic, cardiovascular) as per investigator's discretion
* Known allergies and/or sensitivities to ingredients of Reflex Plus™ or rescue medication
* Regular intake of products that may influence the study outcome, e.g.:

Nutritional Supplement such as vitamin supplements Mineral products, protein, amino acid concentrates Chondroprotective agents such as glucosamine sulfate, chondroitin sulfate, gelatin, hyaluronic acid and methylsulfonylmethane.

Fish oil capsules (omega 3 fatty acid capsules)

* Treatment with cartilage protection products in the last 3 months.
* Treatment (oral ingestion and injection) with steroidal and non-steroidal anti-inflammatory drugs with an exception of the following short-acting NSAID: acetylsalicylic acid, diclofenac, ibuprofen, celecoxib; other analgesics e.g. paracetamol, metamizole and phenazone.
* Cortisone treatment within less than 3 weeks prior to study inclusion.
* Intake of Opioid analgesics.
* Intake of anticoagulants of the coumarin type, such as acenocoumarol and phenprocoumon.
* Simultaneous treatment of osteoarthritis of knee with magnetic therapy, shockwave therapy, acupuncture
* Smokers will be excluded from the study. Occasional smokers willing to abstain smoking during the study can be considered.
* History of drug and alcohol abuse.
* Simultaneous participation in another clinical trial or participation in such within the last 6 weeks.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Reduction from baseline in total score of WOMAC osteoarthritis index at Week 12. | 12 week for protocol A
  To study the change in WOMAC index score from Baseline to Week 12 with respect to: Pain, Stiffness, Physical Function .Total WOMAC score 27 we expect a decrease from baseline WOMAC score in the subjects with knee joint pain.
Reduction from baseline in total score of WOMAC osteoarthritis index at Week 24. | 24 week for protocol B
  To study the change in WOMAC index score from Baseline to Week 24 with respect to: Pain, Stiffness, Physical Function .Total WOMAC score 27 we expect a decrease from baseline WOMAC score in the subjects with knee joint pain.

SECONDARY OUTCOMES:
Reduction in anti-inflammatory markers measured as change from baseline in Serum C reactive protein (CRP) at Week 12. | 12 week for protocol A
  To study the change on anti-inflammatory markers, Serum C reactive protein (CRP) measured from baseline to Week 12.
  C- reactive protein Normal Range is < 5.0 mg/dl which is expected to be raised in subjects with Osteoarthritis.
Reduction of anti-inflammatory markers measured as change from baseline in Serum C reactive protein (CRP) at Week 24. | 24 week for protocol B
  To study the change on anti-inflammatory markers, Serum C reactive protein (CRP) measured from baseline to Week 24.
  C- reactive protein Normal Range is < 5.0 mg/dl which is expected to be raised in subjects with Osteoarthritis.
Increase in joint flexibility measured as change from baseline in axis and range of motion as assess by goniometry at Week 12.baseline in axis and range of motion as assess by goniometry at Week 12 | 12 week for protocol A
  To study the change on joint flexibility measured as change from baseline by goniometry to Week 12.
  Joint Inspection Joint Palpation,Impaired Movement,Axis of Joint,Range of Motion We expect change in range of motion as assessed by goniometry
Increase in joint flexibility measured as change from baseline in axis and range of motion as assess by goniometry at Week 12.baseline in axis and range of motion as assess by goniometry at Week 24 | 24 week for protocol B
  To study the change on joint flexibility measured as change from baseline by goniometry to Week 24.
  Joint Inspection Joint Palpation,Impaired Movement,Axis of Joint,Range of Motion To study the change in MRI for index joint as change from baseline to Week 24.we expect change in range of motion as assessed by goniometry Joint Inspection Joint Palpation,Impaired Movement,Axis of Joint,Range of Motion To study the change in MRI for index joint as change from baseline to Week 24.we expect change in range of motion as assesed by goinometry
Improvement in structure cartilage of knee joint measured as change in MRI analysis from baseline to Week 24. | 24 weeks for protocol B
  To study the effect of Reflex Plus™ on structure of knee joint measured as change in MRI analysis from baseline to Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sachin Dighe, B.A.M.S., Study Director — sachin.d@vediclifesciences.com
Locations (1):
- Mukund Hospital, Mumbai, Maharashtra, India